CLINICAL TRIAL: NCT01761019
Title: A Preliminary, Open Label, Single-arm Study to Determine the Efficacy of Taclonex Topical Suspension as a Supplement to Non-biologic Systemic Therapy
Brief Title: A Study to Determine the Efficacy of Taclonex Topical Suspension as a Supplement to Non-biologic Systemic Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Principal Investigator, Laura Ferris, MD, PhD, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO12100308
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-08

CONDITIONS: Psoriasis
Keywords: psoriasis; Taclonex; Acitretin; Methotrexate
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Taclonex topical suspension (Other): Taclonex topical suspension will be used daily to affected areas of skin with psoriasis for 12 weeks
  Interventions: Drug: Taclonex Topical Suspension

INTERVENTIONS:
Drug: Taclonex Topical Suspension — topical medication for psoriasis

SUMMARY:
Oral therapies for psoriasis, including methotrexate and acitretin, are often less effective when used as monotherapy (without other oral medicines or creams) than are newer biologic injected drugs. However, these oral medications are also less expensive than biologic agents and may be safer for use in some patients. The purpose of this study is to determine if adding a topical psoriasis medicine, calcipotriene/betamethasone topical suspension (Taclonex topical suspension), will improve the severity of psoriasis in patients already on methotrexate or acitretin and to determine if adding this topical suspension will reduce the desire of such patients to switch to a biologic agent to treat their psoriasis.

DETAILED DESCRIPTION:
Many patients with mild psoriasis are able to control disease symptoms with topical medications alone. There are a variety of topical options available, including corticosteroids, synthetic vitamin D3, vitamin A, coal tar, salicylic acid and a number of other products of varying efficacy. The combination topical suspension of calcipotriene 0.005% and betamethasone dipropionate 0.064% is a first-line treatment for moderate to severe psoriasis vulgaris and is FDA approved for use on the skin and scalp in adults 18 years and older. This treatment combines the pharmacological effects of calcipotriene hydrate as a synthetic vitamin D3 analog and betamethasone dipropionate as a synthetic corticosteroid. It is well tolerated and has a low rate of adverse events according to pooled safety data from 2700 patients who have used a calcipotriene/betamethasone combination in clinical trials. Calcipotriene/betamethasone topical suspension has also been shown to have a positive impact on patient quality of life, as seen in clinical trials utilizing patient reported outcomes such as the Dermatology Life Quality Index (DLQI) and Psoriasis Disability Index.

Calcipotriene/betamethasone topical suspension is a therapy commonly used to treat patients with mild to moderate psoriasis. Currently, there have been no formal trials studying the efficacy of calcipotriene/betamethasone topical suspension used in conjunction with methotrexate or acitretin. In order to better understand the effectiveness of this treatment combination, we conducted a preliminary, open label, single arm prospective study to determine the benefit of adding betamethasone-calcipotriene topical suspension to ongoing systemic psoriasis therapy in subjects who do not have complete clearance of psoriasis on a single systemic agent alone.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 years and older with stable plaque psoriasis of duration of at least 6 months.
* Subject must be currently using a stable dose, with stable disease severity, of a single non-biologic systemic psoriasis medication (methotrexate or acitretin) for at least 2 months.
* Subject must be planning to continue current systemic agent, and standard of care monitoring for that medication
* All labs required for methotrexate or acitretin will be done according to standard of care.
* If a woman, before entry she must be: Postmenopausal, or practicing a highly effective method of birth control
* Women of childbearing potential must have a negative urine pregnancy test prior to randomization
* Subject must be able and willing to provide written informed consent to participate.

Exclusion Criteria:

* Non-plaque psoriasis (pustular, erythrodermic, or guttate).
* Use of excluded therapies: phototherapy use currently or in the 4 weeks prior to baseline, use of more than 1 systemic therapy in the 2 months prior to baseline, use of topical steroid, tar preparation, or vitamin D analog in the 4 weeks prior to baseline.
* Subjects who are currently taking or have taken in the past 60 days, for any reason, any medication that, in the opinion of the investigator, suppressed the immune response. This may include but is not limited to systemic steroids, azathioprine, cyclosporine, FK506, mycophenolate mofetil, mycophenolic acid, etanercept, adalimumab, infliximab, ustekinumab, cimzia, or any other biologic agent targeted to any cell or cytokine in the immune system.
* Subjects with any use at any time in the past of Taclonex topical suspension or Taclonex ointment
* Subjects who are pregnant, nursing, or plan on becoming pregnant during the course of the study.
* Presence of any unstable medical or psychiatric condition that, in the opinion of the investigator, could impair subject compliance.
* Subject has any active infection within 30 days prior to baseline.
* Known or suspected disorders of calcium metabolism
* Known or suspected severe kidney or liver disease.
* Known or suspected hypersensitivity to component(s) of the investigational products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Ferris, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Department of Dermatology, Falk Clinic, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Ferris LK, Kupetsky E, Houston NA. A Preliminary, Open Label, Single-arm Study of Calcipotriene/Betamethasone Topical Suspension as a Supplement to Non-biologic Systemic Therapy for Psoriasis. J Clin Aesthet Dermatol. 2016 Apr;9(4):33-8. Epub 2016 Apr 1. PMID 27462386
- See also: UPMC Dermatology Clinical Trials — http://www.upmc.com/Services/dermatology/department-of-derm/clinical-trials/Pages/clinical-trials.aspx

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Taclonex Topical Suspension
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Taclonex Topical Suspension
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 51.375 [38 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment
Description: This is score from 0-5 that measures, in the opinion of the study doctor, the severity of psoriasis on a subject, with 5 being most severe and 0 least severe. The change in this score between baseline and week 12 will be measured.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taclonex Topical Suspension
Number analyzed (Participants) | 8
units on a scale | 1.13 (0.35)

2. Secondary Outcome: Body Surface Area
Description: This is a measure of the percentage of the body involved with psoriasis. We will measure the change in percentage of body area involved with psoriasis from baseline to week 12.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of body surface area
Arm/Group | Taclonex Topical Suspension
Number analyzed (Participants) | 8
percentage of body surface area | 0.7 (0.69)

3. Secondary Outcome: Safety
Description: Throughout this study, adverse events and serious adverse events will be collected
Time Frame: 12 weeks
Measure: Number; unit: adverse event
Arm/Group | Taclonex Topical Suspension
Number analyzed (Participants) | 8
adverse event | 1

4. Secondary Outcome: Patient Satisfaction
Description: • Subject satisfaction: We also ask subjects for their level of satisfaction with their current treatment at week 12. They will be given the following options: "very satisfied", "satisfied", "somewhat disappointed" or "very disappointed". For measurement "very satisfied"=4, "satisfied"=3, "somewhat disappointed"=2 and "very disappointed"=1. We will determine the mean satisfaction of all patients at week 12.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taclonex Topical Suspension
Number analyzed (Participants) | 8
units on a scale | 3.63 (0.52)

5. Secondary Outcome: Desire to Change to Another Systemic Therapy
Description: We will measure the difference in percent of subjects who wish to change to another systemic therapy at baseline vs at week 12.
Time Frame: 12 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Taclonex Topical Suspension
Number analyzed (Participants) | 8
Percentage of participants | 0

ADVERSE EVENTS:
Time Frame: 1 year, 9 months.
Arm/Group | Taclonex Topical Suspension
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Taclonex Topical Suspension (N=8)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The greatest limitation of this study was the small sample size. Other study limitations include the open label, non-randomized design and absence of a placebo arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No